CLINICAL TRIAL: NCT00238602
Title: Evaluation of the Cyberknife Precision Radiation Delivery System for Unresectable Malignant Lung Tumors - A Phase I/II Study
Brief Title: Evaluation of Cyberknife Precision Radiation Delivery System for Unresectable Malignant Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUN0008; 78730; LUN0008; NCT00238602
Record Dates: First submitted 2005-10-11; First posted 2005-10-13 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiosurgery

INTERVENTIONS:
Procedure: Stereotactic radiosurgery

SUMMARY:
This study has two primary objectives. The first objective is to determine the maximal tolerated dose (MTD) that can be delivered with stereotactic radiosurgery in patients with inoperable malignant lung tumors. Once the MTD is established, the second objective is to determine the efficacy of radiosurgical ablation of lung tumors in terms of symptoms and radiographic responses.

ELIGIBILITY:
Inclusion Criteria:1.Lung tumor >= 5.0 cm.

2.Age > 18 years,

3.Histologic confirmation of malignancy (primary lung or metastatic tumor)

4.Deemed unresectable either by radiographic criteria (such as direct invasion of the mediastinum, heart, great vessels, or trachea), by virtue of excessive risk to patient, patient refusal to undergo surgery, or prior operative findings.

5.Performance status of 0-2 by Eastern Clinical Oncology Group criteria Exclusion Criteria:1. No chemotherapy within 2 weeks of radiation treatment.

2. Refusal to sign informed consent.

3. Refusal to take a pregnancy test prior to treatment if the patient is a woman with child bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2000-03; Primary Completion 2007-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Maximal tolerated dose (MTD) that can be delivered with stereotactic radiosurgery in patients with inoperable malignant lung tumors
Efficacy of radiosurgical ablation of lung tumors in terms of symptoms and radiographic responses

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Billy W. Loo Jr. M.D. Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States